CLINICAL TRIAL: NCT00140829
Title: Clinical and Genetic Analysis of Autosomal Recessive Forms of Cerebellar Ataxias and Spastic Paraplegias
Brief Title: SPATAX: Clinical and Genetic Analysis of Cerebellar Ataxias and Spastic Paraplegias
Acronym: Spatax
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Institut des Maladies Rares (Unknown); National Research Agency, France (Other); Paris Brain Institute (ICM) (Other)
Responsible Party: Sponsor
Other Study IDs: RBM01-29; DGS2005/003 (Registry Identifier: N° DGS)
Record Dates: First submitted 2005-08-25; First posted 2005-09-01 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cerebellar Ataxias; Spastic Paraplegias
Keywords: Cerebellar ataxias; Spastic paraplegias; Mutations spectrum; Linkage studies; Genetic counselling
MeSH Terms: conditions — Cerebellar Ataxia; Paraplegia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA and LH tubes to be able to extract DNA from blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Cerebellar ataxias (CA) and spastic paraplegias (SP) are genetically and clinically very heterogeneous. More than 40 loci are already known but the number of phenotypes is even greater suggesting further genetic heterogeneity. These progressive disorders are often severe and fatal, due to the absence of specific therapy. The SPATAX network combines the experience of European clinicians and scientists working on these groups of diseases. Over the past year, they have assembled the largest collection of families and achieved a number of tasks (initiation of a clinical and genetic database, distribution of DNA to participating laboratories, mapping of three new loci, and refinement of several loci). In addition to clinicians from Europe and Mediterranean countries, who play a major role in collecting families according to evaluation tools developed and validated by the SPATAX members, the group includes major European laboratories devoted to the elucidation of the molecular basis of these disorders. Each laboratory will centralize all families with a subtype of autosomal recessive (AR) CA (n=116) or SP (n=207) in order to efficiently map and identify the responsible gene(s). Genome-wide scans are already underway in 61 families. Given the expertise of the participants, the researchers expect to map and identify several genes during the course of this project. The spectrum of mutations and phenotype/genotype correlations will be analysed thanks to this unique series of patients with various phenotypes. The knowledge gained will be immediately applicable to patients in terms of improved positive diagnosis, follow-up and appropriate genetic counselling. In the long term, models for genetic entity will be developed in order to understand the pathophysiology and to identify new targets for treatment. The series of patients assembled and the precise knowledge of natural history will facilitate the implantation of therapeutic trials based on rational approaches.

ELIGIBILITY:
Inclusion Criteria:

* Progressive ataxia or paraplegia

Exclusion Criteria:

* Lack of signed informed consent

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: French population
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2004-02-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Characterize clinically the different forms of these diseases | Year 1 to Year 7
  Validation of a new quantitative tool with more sensitive grading scale of cerebellar syndrome, spasticity and their consequences. In one single device, three tests were assessed for hand coordination ( " tapping test ", " peg board test" and " click test "), one test for dysarthria and a final test to quantify walking disorders due to spasticity (distance covered in 5 seconds).
Elucidate the molecular bases of these diseases | through study duration (through study duration (up to 14 years) )
  To elucidate the molecular bases of these diseases (identify the loci/genes involved as well as those that modulate their expression) in order to enable the development of molecular diagnostics, the study of disease mechanisms, the identification of biomarkers and, subsequently, to propose new treatments.
Establish the natural history of spino-cerebellar degeneration | Year 1 to Year 7
  Investigators intended to follow the clinical status of this cohort of patients for 7 years, by assessing the progression of the pathology each year with a neurological exam

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Dürr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Alessandro Filla, MD, PhD, Principal Investigator — Federico II University; André Mégarbané, MD, Principal Investigator — Université Saint-Joseph; Ali Benomar, MD, PhD, Principal Investigator — CHU de Rabat; Christophe Verny, MD, Principal Investigator — University Hospital, Angers; Didier Hannequin, MD, PhD, Principal Investigator — Hôpitaux de Rouen; Diana Rodriguez, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Enrico Bertini, MD, Principal Investigator — Università de Roma; François Tison, MD, PhD, Principal Investigator — Hôpitaux de Bordeaux; Jorgen E Nielsen, MD, PhD, Principal Investigator — The Panum Institute; Mustapha Salih, MD, Principal Investigator — College of Medicine and KKUH; Miriem Tazir, MD, PhD, Principal Investigator — Université d'Alger; Nicholas W Wood, MD, PhD, Principal Investigator — Institute of Neurology; Odile Boespflug-Tanguy, MD, PhD, Principal Investigator — Hôpitaux de Clermont-Ferrand; Jean-Philippe Azulay, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Marseille; Paula Coutinho, MD, PhD, Principal Investigator — Universidade do Porto; Pierre Labauge, MD, PhD, Principal Investigator — Hôpitaux de Nîmes; Pierre Pollak, MD, PhD, Principal Investigator — Hôpitaux de Grenoble; Thomas T Warner, MD, PhD, Principal Investigator — University College, London; Alexander Lossos, MD, Principal Investigator — Hadassah-Hebrew University Hospital; Cyril Goizet, MD, PhD, Principal Investigator — Hôpital Pellegrin; Patrick Calvas, MD, PhD, Principal Investigator — Hôpital Purpan; Berry Kremer, MD, Principal Investigator — Radboud University Medical Center; Vladimir Kostic, MD, Principal Investigator — Clinical Centre of Serbia; Chokri Mhiri, MD, Principal Investigator — Hôpital Habib Bourguiba; Massimo Pandolfo, MD, PhD, Principal Investigator — Université Libre de Bruxelles - Hôpital Erasme; Jorge Sequeiros, MD, PhD, Principal Investigator — Universidade do Porto; Chantal ME Tallaksen, MD, PhD, Principal Investigator — Ullevaal University Hospital
Locations (27):
- CHU Mustapha, Algiers, Algeria
- Université Libre de Bruxelles - Hôpital Erasme, Brussels, Belgium
- The Panum Institute, Copenhagen, Denmark
- France (10):
  - CHU d'Angers, Angers
  - Hôpital Pellegrin, Bordeaux
  - Hôpitaux de Clermont-Ferrand, Clermont-Ferrand
  - CHU, Grenoble
  - Hôpital de la Timone, Marseille
  - Hôpital Carémeau, Nîmes
  - Hôpital Armand Trousseau, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse
- Hadassah-Hebrew University Hospital, Jerusalem, Israel
- Italy (2):
  - Dipartimento Di Scienze Neurologiche, Napoli
  - Molecular Medicine and Department of Neurosciences, Roma
- Université Saint-Joseph, Beirut, Lebanon
- CHU de Rabat, Rabat, Morocco
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Ullevål University Hospital, Oslo, Norway
- Portugal (2):
  - University of Porto, Porto
  - Hospital San Sebastião, Santa Maria da Feira
- King Khalid University Hospital, Riyadh, Saudi Arabia
- Clinical Centre of Serbia, Belgrade, Serbia
- Hôpital Habib Bourguiba, Sfax, Tunisia
- United Kingdom (2):
  - Royal Free and University College Medical School, London
  - The National Hospital, London

REFERENCES:
- [Background] Moreira MC, Klur S, Watanabe M, Nemeth AH, Le Ber I, Moniz JC, Tranchant C, Aubourg P, Tazir M, Schols L, Pandolfo M, Schulz JB, Pouget J, Calvas P, Shizuka-Ikeda M, Shoji M, Tanaka M, Izatt L, Shaw CE, M'Zahem A, Dunne E, Bomont P, Benhassine T, Bouslam N, Stevanin G, Brice A, Guimaraes J, Mendonca P, Barbot C, Coutinho P, Sequeiros J, Durr A, Warter JM, Koenig M. Senataxin, the ortholog of a yeast RNA helicase, is mutant in ataxia-ocular apraxia 2. Nat Genet. 2004 Mar;36(3):225-7. doi: 10.1038/ng1303. Epub 2004 Feb 8. PMID 14770181
- [Background] Le Ber I, Bouslam N, Rivaud-Pechoux S, Guimaraes J, Benomar A, Chamayou C, Goizet C, Moreira MC, Klur S, Yahyaoui M, Agid Y, Koenig M, Stevanin G, Brice A, Durr A. Frequency and phenotypic spectrum of ataxia with oculomotor apraxia 2: a clinical and genetic study in 18 patients. Brain. 2004 Apr;127(Pt 4):759-67. doi: 10.1093/brain/awh080. Epub 2004 Jan 21. PMID 14736755
- [Background] Le Ber I, Moreira MC, Rivaud-Pechoux S, Chamayou C, Ochsner F, Kuntzer T, Tardieu M, Said G, Habert MO, Demarquay G, Tannier C, Beis JM, Brice A, Koenig M, Durr A. Cerebellar ataxia with oculomotor apraxia type 1: clinical and genetic studies. Brain. 2003 Dec;126(Pt 12):2761-72. doi: 10.1093/brain/awg283. Epub 2003 Sep 23. PMID 14506070
- [Background] Le Ber I, Camuzat A, Castelnovo G, Azulay JP, Genton P, Gastaut JL, Broglin D, Labauge P, Brice A, Durr A. Prevalence of dentatorubral-pallidoluysian atrophy in a large series of white patients with cerebellar ataxia. Arch Neurol. 2003 Aug;60(8):1097-9. doi: 10.1001/archneur.60.8.1097. PMID 12925365
- [Background] Bouslam N, Benomar A, Azzedine H, Bouhouche A, Namekawa M, Klebe S, Charon C, Durr A, Ruberg M, Brice A, Yahyaoui M, Stevanin G. Mapping of a new form of pure autosomal recessive spastic paraplegia (SPG28). Ann Neurol. 2005 Apr;57(4):567-71. doi: 10.1002/ana.20416. PMID 15786464
- [Background] Durr A, Camuzat A, Colin E, Tallaksen C, Hannequin D, Coutinho P, Fontaine B, Rossi A, Gil R, Rousselle C, Ruberg M, Stevanin G, Brice A. Atlastin1 mutations are frequent in young-onset autosomal dominant spastic paraplegia. Arch Neurol. 2004 Dec;61(12):1867-72. doi: 10.1001/archneur.61.12.1867. PMID 15596607
- [Background] Stevanin G, Durr A, Dussert C, Penet C, Brice A. Mutations in the FGF14 gene are not a major cause of spinocerebellar ataxia in Caucasians. Neurology. 2004 Sep 14;63(5):936. doi: 10.1212/01.wnl.0000137020.30604.1e. No abstract available. PMID 15365159
- [Background] Stevanin G, Hahn V, Lohmann E, Bouslam N, Gouttard M, Soumphonphakdy C, Welter ML, Ollagnon-Roman E, Lemainque A, Ruberg M, Brice A, Durr A. Mutation in the catalytic domain of protein kinase C gamma and extension of the phenotype associated with spinocerebellar ataxia type 14. Arch Neurol. 2004 Aug;61(8):1242-8. doi: 10.1001/archneur.61.8.1242. PMID 15313841
- [Background] Stevanin G, Bouslam N, Thobois S, Azzedine H, Ravaux L, Boland A, Schalling M, Broussolle E, Durr A, Brice A. Spinocerebellar ataxia with sensory neuropathy (SCA25) maps to chromosome 2p. Ann Neurol. 2004 Jan;55(1):97-104. doi: 10.1002/ana.10798. PMID 14705117
- [Background] Tallaksen CM, Guichart-Gomez E, Verpillat P, Hahn-Barma V, Ruberg M, Fontaine B, Brice A, Dubois B, Durr A. Subtle cognitive impairment but no dementia in patients with spastin mutations. Arch Neurol. 2003 Aug;60(8):1113-8. doi: 10.1001/archneur.60.8.1113. PMID 12925368
- [Background] Fernet M, Gribaa M, Salih MA, Seidahmed MZ, Hall J, Koenig M. Identification and functional consequences of a novel MRE11 mutation affecting 10 Saudi Arabian patients with the ataxia telangiectasia-like disorder. Hum Mol Genet. 2005 Jan 15;14(2):307-18. doi: 10.1093/hmg/ddi027. Epub 2004 Dec 1. PMID 15574463
- [Background] Stevanin G, Durr A, Benammar N, Brice A. Spinocerebellar ataxia with mental retardation (SCA13). Cerebellum. 2005;4(1):43-6. doi: 10.1080/14734220510007923. PMID 15895558
- [Background] Stevanin G, Broussolle E, Streichenberger N, Kopp N, Brice A, Durr A. Spinocerebellar ataxia with sensory neuropathy (SCA25). Cerebellum. 2005;4(1):58-61. doi: 10.1080/14734220510007932. PMID 15895562
- [Background] Klebe S, Durr A, Rentschler A, Hahn-Barma V, Abele M, Bouslam N, Schols L, Jedynak P, Forlani S, Denis E, Dussert C, Agid Y, Bauer P, Globas C, Wullner U, Brice A, Riess O, Stevanin G. New mutations in protein kinase Cgamma associated with spinocerebellar ataxia type 14. Ann Neurol. 2005 Nov;58(5):720-9. doi: 10.1002/ana.20628. PMID 16193476
- [Background] Latouche M, Fragner P, Martin E, El Hachimi KH, Zander C, Sittler A, Ruberg M, Brice A, Stevanin G. Polyglutamine and polyalanine expansions in ataxin7 result in different types of aggregation and levels of toxicity. Mol Cell Neurosci. 2006 Mar;31(3):438-45. doi: 10.1016/j.mcn.2005.10.013. Epub 2005 Dec 1. PMID 16325416
- [Background] Namekawa M, Ribai P, Nelson I, Forlani S, Fellmann F, Goizet C, Depienne C, Stevanin G, Ruberg M, Durr A, Brice A. SPG3A is the most frequent cause of hereditary spastic paraplegia with onset before age 10 years. Neurology. 2006 Jan 10;66(1):112-4. doi: 10.1212/01.wnl.0000191390.20564.8e. PMID 16401858
- [Background] van de Warrenburg BP, Hendriks H, Durr A, van Zuijlen MC, Stevanin G, Camuzat A, Sinke RJ, Brice A, Kremer BP. Age at onset variance analysis in spinocerebellar ataxias: a study in a Dutch-French cohort. Ann Neurol. 2005 Apr;57(4):505-12. doi: 10.1002/ana.20424. PMID 15747371
- [Background] Biancalana V, Toft M, Le Ber I, Tison F, Scherrer E, Thibodeau S, Mandel JL, Brice A, Farrer MJ, Durr A. FMR1 premutations associated with fragile X-associated tremor/ataxia syndrome in multiple system atrophy. Arch Neurol. 2005 Jun;62(6):962-6. doi: 10.1001/archneur.62.6.962. PMID 15956167
- [Background] Ribaï P, Stevanin G, Trefouret S, Nelson I, Soumphonphakdy C, Pouget J, Dürr A, Brice A. Extension of the SPG26 phenotype in a Spanish family and refinement of its locus on chromosome 12. Eletter, Journal of Medical Genetics 42(1):80-82, 2005.
- [Background] Elleuch N, Depienne C, Benomar A, Hernandez AM, Ferrer X, Fontaine B, Grid D, Tallaksen CM, Zemmouri R, Stevanin G, Durr A, Brice A. Mutation analysis of the paraplegin gene (SPG7) in patients with hereditary spastic paraplegia. Neurology. 2006 Mar 14;66(5):654-9. doi: 10.1212/01.wnl.0000201185.91110.15. PMID 16534102
- [Background] Le Ber I, Rivaud-Pechoux S, Brice A, Durr A. [Autosomal recessive cerebellar ataxias with oculomotor apraxia]. Rev Neurol (Paris). 2006 Feb;162(2):177-84. doi: 10.1016/s0035-3787(06)74997-9. French. PMID 16518257
- [Background] Namekawa M, Nelson I, Ribai P, Durr A, Denis E, Stevanin G, Ruberg M, Brice A. A founder effect and mutational hot spots may contribute to the most frequent mutations in the SPG3A gene. Neurogenetics. 2006 May;7(2):131-2. doi: 10.1007/s10048-006-0028-2. Epub 2006 Apr 13. No abstract available. PMID 16612642
- [Background] Lossos A, Stevanin G, Meiner V, Argov Z, Bouslam N, Newman JP, Gomori JM, Klebe S, Lerer I, Elleuch N, Silverstein S, Durr A, Abramsky O, Ben-Nariah Z, Brice A. Hereditary spastic paraplegia with thin corpus callosum: reduction of the SPG11 interval and evidence for further genetic heterogeneity. Arch Neurol. 2006 May;63(5):756-60. doi: 10.1001/archneur.63.5.756. PMID 16682547
- [Background] Klebe S, Azzedine H, Durr A, Bastien P, Bouslam N, Elleuch N, Forlani S, Charon C, Koenig M, Melki J, Brice A, Stevanin G. Autosomal recessive spastic paraplegia (SPG30) with mild ataxia and sensory neuropathy maps to chromosome 2q37.3. Brain. 2006 Jun;129(Pt 6):1456-62. doi: 10.1093/brain/awl012. Epub 2006 Jan 24. PMID 16434418
- [Background] Ribai P, Stevanin G, Bouslam N, Pontier B, Nelson I, Fontaine B, Dussert C, Charon C, Durr A, Brice A. A new phenotype linked to SPG27 and refinement of the critical region on chromosome. J Neurol. 2006 Jun;253(6):714-9. doi: 10.1007/s00415-006-0094-2. Epub 2006 Mar 6. PMID 16511635
- [Background] Le Ber I, Clot F, Vercueil L, Camuzat A, Viemont M, Benamar N, De Liege P, Ouvrard-Hernandez AM, Pollak P, Stevanin G, Brice A, Durr A. Predominant dystonia with marked cerebellar atrophy: a rare phenotype in familial dystonia. Neurology. 2006 Nov 28;67(10):1769-73. doi: 10.1212/01.wnl.0000244484.60489.50. PMID 17130408
- [Background] Stevanin G, Montagna G, Azzedine H, Valente EM, Durr A, Scarano V, Bouslam N, Cassandrini D, Denora PS, Criscuolo C, Belarbi S, Orlacchio A, Jonveaux P, Silvestri G, Hernandez AM, De Michele G, Tazir M, Mariotti C, Brockmann K, Malandrini A, van der Knapp MS, Neri M, Tonekaboni H, Melone MA, Tessa A, Dotti MT, Tosetti M, Pauri F, Federico A, Casali C, Cruz VT, Loureiro JL, Zara F, Forlani S, Bertini E, Coutinho P, Filla A, Brice A, Santorelli FM. Spastic paraplegia with thin corpus callosum: description of 20 new families, refinement of the SPG11 locus, candidate gene analysis and evidence of genetic heterogeneity. Neurogenetics. 2006 Jul;7(3):149-56. doi: 10.1007/s10048-006-0044-2. Epub 2006 May 13. PMID 16699786
- [Background] Klebe S, Lacour A, Durr A, Stojkovic T, Depienne C, Forlani S, Poea-Guyon S, Vuillaume I, Sablonniere B, Vermersch P, Brice A, Stevanin G. NIPA1 (SPG6) mutations are a rare cause of autosomal dominant spastic paraplegia in Europe. Neurogenetics. 2007 Apr;8(2):155-7. doi: 10.1007/s10048-006-0074-9. Epub 2007 Jan 5. No abstract available. PMID 17205300
- [Background] Bouslam N, Bouhouche A, Benomar A, Hanein S, Klebe S, Azzedine H, Di Giandomenico S, Boland-Auge A, Santorelli FM, Durr A, Brice A, Yahyaoui M, Stevanin G. A novel locus for autosomal recessive spastic ataxia on chromosome 17p. Hum Genet. 2007 May;121(3-4):413-20. doi: 10.1007/s00439-007-0328-0. Epub 2007 Feb 2. PMID 17273843
- [Background] Stevanin G, Santorelli FM, Azzedine H, Coutinho P, Chomilier J, Denora PS, Martin E, Ouvrard-Hernandez AM, Tessa A, Bouslam N, Lossos A, Charles P, Loureiro JL, Elleuch N, Confavreux C, Cruz VT, Ruberg M, Leguern E, Grid D, Tazir M, Fontaine B, Filla A, Bertini E, Durr A, Brice A. Mutations in SPG11, encoding spatacsin, are a major cause of spastic paraplegia with thin corpus callosum. Nat Genet. 2007 Mar;39(3):366-72. doi: 10.1038/ng1980. Epub 2007 Feb 18. PMID 17322883
- [Background] Latouche M, Lasbleiz C, Martin E, Monnier V, Debeir T, Mouatt-Prigent A, Muriel MP, Morel L, Ruberg M, Brice A, Stevanin G, Tricoire H. A conditional pan-neuronal Drosophila model of spinocerebellar ataxia 7 with a reversible adult phenotype suitable for identifying modifier genes. J Neurosci. 2007 Mar 7;27(10):2483-92. doi: 10.1523/JNEUROSCI.5453-06.2007. PMID 17344386
- [Background] Klebe S, Durr A, Bouslam N, Grid D, Paternotte C, Depienne C, Hanein S, Bouhouche A, Elleuch N, Azzedine H, Poea-Guyon S, Forlani S, Denis E, Charon C, Hazan J, Brice A, Stevanin G. Spastic paraplegia 5: Locus refinement, candidate gene analysis and clinical description. Am J Med Genet B Neuropsychiatr Genet. 2007 Oct 5;144B(7):854-61. doi: 10.1002/ajmg.b.30518. PMID 17503452
- [Background] Stevanin G, Paternotte C, Coutinho P, Klebe S, Elleuch N, Loureiro JL, Denis E, Cruz VT, Durr A, Prud'homme JF, Weissenbach J, Brice A, Hazan J. A new locus for autosomal recessive spastic paraplegia (SPG32) on chromosome 14q12-q21. Neurology. 2007 May 22;68(21):1837-40. doi: 10.1212/01.wnl.0000262043.53386.22. PMID 17515546
- [Background] Namekawa M, Muriel MP, Janer A, Latouche M, Dauphin A, Debeir T, Martin E, Duyckaerts C, Prigent A, Depienne C, Sittler A, Brice A, Ruberg M. Mutations in the SPG3A gene encoding the GTPase atlastin interfere with vesicle trafficking in the ER/Golgi interface and Golgi morphogenesis. Mol Cell Neurosci. 2007 May;35(1):1-13. doi: 10.1016/j.mcn.2007.01.012. Epub 2007 Jan 26. PMID 17321752
- [Background] Stevanin G, Azzedine H, Denora P, Boukhris A, Tazir M, Lossos A, Rosa AL, Lerer I, Hamri A, Alegria P, Loureiro J, Tada M, Hannequin D, Anheim M, Goizet C, Gonzalez-Martinez V, Le Ber I, Forlani S, Iwabuchi K, Meiner V, Uyanik G, Erichsen AK, Feki I, Pasquier F, Belarbi S, Cruz VT, Depienne C, Truchetto J, Garrigues G, Tallaksen C, Tranchant C, Nishizawa M, Vale J, Coutinho P, Santorelli FM, Mhiri C, Brice A, Durr A; SPATAX consortium. Mutations in SPG11 are frequent in autosomal recessive spastic paraplegia with thin corpus callosum, cognitive decline and lower motor neuron degeneration. Brain. 2008 Mar;131(Pt 3):772-84. doi: 10.1093/brain/awm293. Epub 2007 Dec 13. PMID 18079167
- [Background] Boukhris A, Feki I, Denis E, Miladi MI, Brice A, Mhiri C, Stevanin G. Spastic paraplegia 15: linkage and clinical description of three Tunisian families. Mov Disord. 2008 Feb 15;23(3):429-33. doi: 10.1002/mds.21848. PMID 18098276
- [Background] Boukhris A, Stevanin G, Feki I, Denis E, Elleuch N, Miladi MI, Truchetto J, Denora P, Belal S, Mhiri C, Brice A. Hereditary spastic paraplegia with mental impairment and thin corpus callosum in Tunisia: SPG11, SPG15, and further genetic heterogeneity. Arch Neurol. 2008 Mar;65(3):393-402. doi: 10.1001/archneur.65.3.393. PMID 18332254
- [Background] Hanein S, Martin E, Boukhris A, Byrne P, Goizet C, Hamri A, Benomar A, Lossos A, Denora P, Fernandez J, Elleuch N, Forlani S, Durr A, Feki I, Hutchinson M, Santorelli FM, Mhiri C, Brice A, Stevanin G. Identification of the SPG15 gene, encoding spastizin, as a frequent cause of complicated autosomal-recessive spastic paraplegia, including Kjellin syndrome. Am J Hum Genet. 2008 Apr;82(4):992-1002. doi: 10.1016/j.ajhg.2008.03.004. PMID 18394578
- [Background] Denora PS, Schlesinger D, Casali C, Kok F, Tessa A, Boukhris A, Azzedine H, Dotti MT, Bruno C, Truchetto J, Biancheri R, Fedirko E, Di Rocco M, Bueno C, Malandrini A, Battini R, Sickl E, de Leva MF, Boespflug-Tanguy O, Silvestri G, Simonati A, Said E, Ferbert A, Criscuolo C, Heinimann K, Modoni A, Weber P, Palmeri S, Plasilova M, Pauri F, Cassandrini D, Battisti C, Pini A, Tosetti M, Hauser E, Masciullo M, Di Fabio R, Piccolo F, Denis E, Cioni G, Massa R, Della Giustina E, Calabrese O, Melone MA, De Michele G, Federico A, Bertini E, Durr A, Brockmann K, van der Knaap MS, Zatz M, Filla A, Brice A, Stevanin G, Santorelli FM. Screening of ARHSP-TCC patients expands the spectrum of SPG11 mutations and includes a large scale gene deletion. Hum Mutat. 2009 Mar;30(3):E500-19. doi: 10.1002/humu.20945. PMID 19105190
- [Background] Denora PS, Muglia M, Casali C, Truchetto J, Silvestri G, Messina D, Boukrhis A, Magariello A, Modoni A, Masciullo M, Malandrini A, Morelli M, de Leva MF, Villanova M, Giugni E, Citrigno L, Rizza T, Federico A, Pierallini A, Quattrone A, Filla A, Brice A, Stevanin G, Santorelli FM. Spastic paraplegia with thinning of the corpus callosum and white matter abnormalities: further mutations and relative frequency in ZFYVE26/SPG15 in the Italian population. J Neurol Sci. 2009 Feb 15;277(1-2):22-5. doi: 10.1016/j.jns.2008.09.039. Epub 2008 Dec 13. PMID 19084844
- [Background] Boukhris A, Stevanin G, Feki I, Denora P, Elleuch N, Miladi MI, Goizet C, Truchetto J, Belal S, Brice A, Mhiri C. Tunisian hereditary spastic paraplegias: clinical variability supported by genetic heterogeneity. Clin Genet. 2009 Jun;75(6):527-36. doi: 10.1111/j.1399-0004.2009.01176.x. Epub 2009 May 5. PMID 19438933
- [Background] Anheim M, Lagier-Tourenne C, Stevanin G, Fleury M, Durr A, Namer IJ, Denora P, Brice A, Mandel JL, Koenig M, Tranchant C. SPG11 spastic paraplegia. A new cause of juvenile parkinsonism. J Neurol. 2009 Jan;256(1):104-8. doi: 10.1007/s00415-009-0083-3. Epub 2009 Feb 9. PMID 19224311
- [Background] Goizet C, Boukhris A, Durr A, Beetz C, Truchetto J, Tesson C, Tsaousidou M, Forlani S, Guyant-Marechal L, Fontaine B, Guimaraes J, Isidor B, Chazouilleres O, Wendum D, Grid D, Chevy F, Chinnery PF, Coutinho P, Azulay JP, Feki I, Mochel F, Wolf C, Mhiri C, Crosby A, Brice A, Stevanin G. CYP7B1 mutations in pure and complex forms of hereditary spastic paraplegia type 5. Brain. 2009 Jun;132(Pt 6):1589-600. doi: 10.1093/brain/awp073. Epub 2009 May 12. PMID 19439420
- [Background] Goizet C, Boukhris A, Maltete D, Guyant-Marechal L, Truchetto J, Mundwiller E, Hanein S, Jonveaux P, Roelens F, Loureiro J, Godet E, Forlani S, Melki J, Auer-Grumbach M, Fernandez JC, Martin-Hardy P, Sibon I, Sole G, Orignac I, Mhiri C, Coutinho P, Durr A, Brice A, Stevanin G. SPG15 is the second most common cause of hereditary spastic paraplegia with thin corpus callosum. Neurology. 2009 Oct 6;73(14):1111-9. doi: 10.1212/WNL.0b013e3181bacf59. PMID 19805727
- [Background] Anheim M, Monga B, Fleury M, Charles P, Barbot C, Salih M, Delaunoy JP, Fritsch M, Arning L, Synofzik M, Schols L, Sequeiros J, Goizet C, Marelli C, Le Ber I, Koht J, Gazulla J, De Bleecker J, Mukhtar M, Drouot N, Ali-Pacha L, Benhassine T, Chbicheb M, M'Zahem A, Hamri A, Chabrol B, Pouget J, Murphy R, Watanabe M, Coutinho P, Tazir M, Durr A, Brice A, Tranchant C, Koenig M. Ataxia with oculomotor apraxia type 2: clinical, biological and genotype/phenotype correlation study of a cohort of 90 patients. Brain. 2009 Oct;132(Pt 10):2688-98. doi: 10.1093/brain/awp211. Epub 2009 Aug 20. PMID 19696032
- See also: Related Info — http://www.inserm.fr